CLINICAL TRIAL: NCT05565573
Title: The Therapeutic Effect of Medroxyprogesterone Acetate vs. LNG-IUS in Early-stage Endometrioid Carcinoma
Brief Title: Medroxyprogesterone Acetate vs LNG-IUS in Early-stage Endometrioid Carcinoma and Atypical Hyperplasia Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hua Li (Other)
Responsible Party: Sponsor-Investigator, Hua Li, Department of Obstetrics and Gynecology, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LH0930
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Fertility Sparing
MeSH Terms: interventions — Medroxyprogesterone Acetate; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medroxyprogesterone acetate (Experimental): Administered MPA at a dosage of 500 mg/d concurrently
  Interventions: Drug: Medroxyprogesterone Acetate 500 MG Oral Tablet
- LNG-IUS (Experimental): Go through LNG-IUS insertion
  Interventions: Device: Levonorgestrel-Releasing Intrauterine System

INTERVENTIONS:
Drug: Medroxyprogesterone Acetate 500 MG Oral Tablet — 500mg/ Pfizer Active ingredient: Medroxyprogesterone Acetate At a dosage of 500 mg/day
  Other Names: MPA
  Arms: Medroxyprogesterone acetate
Device: Levonorgestrel-Releasing Intrauterine System — Uterine cavity insertion
  Other Names: LNG-IUS, 52-mg LNG-IUS，Mirena
  Arms: LNG-IUS

SUMMARY:
In modern society, endometrial cancer (EC) and atypical hyperplasia is the most frequent desease which can affect the fertility of young patients. For young patients, there is a growing need to treat tumors and fertility sparing. Advaced studies have confirmed thatfertility preservation therapy has better tumor and pregnancy outcomes in specific patients with early gynecological tumors. Clinically, evidence-based guidelines are urgently needed to guide the screening and treatment of women who are suitable for fertility preservation. Fertility-sparing treatment predominantly involves the use of oral progestins and levonorgestrel-releasing intrauterine devices, which have been shown to be feasible and safe in women with early stage EC and minimal or no myometrial invasion. However, data on the efficacy and safety of conservative management strategies are primarily based on retrospective studies.The present study aims to compared the therapeutic effect of Medroxyprogesterone acetate (MPA) and Levonorgestrel-releasing intrauterine system (LNG-IUS) in early-stage endometrioid carcinoma and atypical hyperplasia patients

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 45 years old;
2. Diagnostic curettage pathology is highly differentiated endometrioid adenocarcinoma;
3. pelvic augmentation MRI or / and vaginal color ultrasound Doppler examination, tumor confined endometrium;
4. No suspicious metastatic lesions;
5. Endometrial pathological tissue specimens with strong positive expression of estrogen and progesterone receptors;
6. Blood CA125 is normal;
7. no progesterone therapy and contraindications to pregnancy;
8. The patient himself has a strong desire to preserve fertility, and the patient should fully understand that fertility preservation treatment is not the standard treatment method;
9. Conditional acceptance of close follow-up.

Exclusion Criteria:

1. type II endometrial cancer;
2. Patients with abnormal liver and kidney function and other contraindications to progesterone therapy;
3. Other parts of the body are concurrent or successively complicated by other malignant tumors;
4. The patient and his/her family are unable to sign the informed consent form for any reason;
5. Unconditional follow-up.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 24-week
  The 24-week CR rate will be calculated in two groups.

SECONDARY OUTCOMES:
Time to achieve complete response | From date of randomization until the date of CR, assessed up to 24 weeks
  The median CR time will be calculated in two groups
The pregnancy rate | Up to 2 years after the treatment
  Rate of fertility outcomes
The live-birth rate | Up to 2 years after the treatment
  Rate of fertility outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Hua Li, Ph.D, Study Chair — Beijing Chao Yang Hospital
Locations (1):
- Bei Jing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No